CLINICAL TRIAL: NCT02565485
Title: Pulse Pressure-guided IV Fluid Preload to Prevent Post-epidural Fetal Heart Rate (FHR) Changes: a Randomized Controlled Trial
Brief Title: Pulse Pressure and Post-epidural Fetal Heart Rate Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Edward Chien, MD, Professor, Reproductive Biology, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB15-00366
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Fetus or Neonate Affected by Maternal Epidural Anesthesia During Labor and Delivery
Keywords: pulse pressure; fetal heart rate; epidural analgesia; hypotension; preload; fluid bolus; central hypovolemia
MeSH Terms: conditions — Hypotension | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard IV Preload (No Intervention): Patients in this arm will receive 500mL of Lactated Ringer's solution, which is the standard IV fluid preload used on Labor and Delivery at MetroHealth Medical Center
- Volume Replacement IV Preload (Experimental): Patients in this arm will receive 1500mL of Lactated Ringer's solution
  Interventions: Drug: Lactated Ringer's

INTERVENTIONS:
Drug: Lactated Ringer's — 1500 cc of IV Fluid (crystalloid) used for preload prior to epidural administration in the treatment arm. Control arm receives 500 cc.
  Other Names: Ringer's Lactate
  Arms: Volume Replacement IV Preload

SUMMARY:
Epidural anesthesia, the most common method of pain control in labor, can contribute to alterations in maternal blood pressure and/or fetal heart rate changes. As a result, the administration of an IV fluid bolus ("preload") is standard prior to epidural placement. However, the optimal volume of preload is unknown and no clinical trials have evaluated a risk-factor based approach to dosing. Studies in the critical care, trauma, and obstetric literature have suggested that a narrow pulse pressure (difference between systolic and diastolic blood pressures) is a marker of reduced intravascular volume status and may identify women at a higher risk for new onset fetal heart rate changes after epidural placement. Therefore, the purpose of this study is to assess if an increased IV fluid preload bolus among women with a narrow pulse pressure reduces the risk of new onset fetal heart rate changes after epidural placement.

DETAILED DESCRIPTION:
Objective:

To assess the efficacy of increased IV fluid preload for the prevention of post-epidural FHR changes in women with narrow pulse pressure

Hypothesis:

In individual with narrow pulse pressure, an increased IV fluid bolus will reduce the rate of post-epidural FHR changes.

Background:

In contemporary obstetric practice, regional anesthesia is the most commonly utilized method for pain management in labor. Compared with no anesthesia, neuraxial techniques have been associated with an increased risk of maternal hypotension, operative vaginal delivery, maternal fever, and cesarean delivery for fetal distress. Following the initial dosing of regional anesthesia, maternal hypotension and FHR abnormalities occur with reported frequencies of 5-18% and 6-30% respectively.

Neuraxial anesthesia can induce a sympathetic blockade, which results in decreased maternal systemic vascular resistance and venous return. These alterations in the maternal hemodynamic profile impact maternal blood pressure, uteroplacental blood flow and fetal perfusion, and may contribute to maternal hypotension and changes in the FHR after initiation of regional anesthesia. Importantly, these hemodynamic changes generally occur in the setting of a constant maternal intravascular volume. Given that the uteroplacental circulation has limited capacity for autoregulation, uterine perfusion is sensitive to changes in both maternal blood pressure and venous return. This physiology represents the basis for the administration of an intravenous (IV) bolus prior to or during the placement of regional anesthesia .

While maternal hypotension and FHR changes after neuraxial anesthesia are common occurrences, limited information on maternal and fetal characteristics or risk factors has been published. A recent retrospective cohort study by Miller et al. reported that a narrow maternal pulse pressure was a risk factor for post-epidural FHR changes. In this cohort study, women with an admission pulse pressure < 45, compared with pulse pressure > 45, had a marked increase in the risk of post-epidural FHR changes (27% vs 6%, p < 0.001, OR 5.6 [2.1-14.3], aOR 28.9 [3.8-221.4]). Interestingly, the incidence of maternal hypotension was not different between the two pulse pressure groups (21% vs 25%, p=0.49), suggesting that fetal perfusion is sensitive to the reduced venous return associated with increased venous capacitance related to reduced sympathetic tone. Further supporting this premise, a study by Vricella et al. demonstrated an increased rate of post-epidural maternal hypotension, vasopressor support and FHR changes in women with severe preeclampsia, a clinical state of volume contraction, compared with normotensive controls. The authors concluded that the vasoconstriction and intravascular depletion central to the syndrome of severe preeclampsia make this subset of women vulnerable to post-epidural hemodynamic changes and that administration of a standard IV fluid bolus may not adequately compensate for increased venous capacitance.

Data from the critical care and trauma literature further support the use of pulse pressure as a marker of hypovolemia. Conventional static indicators of cardiac preload, such as central venous pressure (CVP) or pulmonary capillary wedge pressure (PCWP), are poor predictors of "volume responsiveness", which is the cardiovascular response (i.e. changes in preload) to intravascular volume expansion with IV fluid. However, dynamic parameters such as variation in pulse pressure or stroke volume, are highly predictive of volume responsiveness. While data on pulse pressure variation are primarily derived from non-pregnant, mechanically ventilated individuals, a small case series demonstrated that pulse pressure variation accurately reflects volume responsiveness in pregnant women undergoing cesarean delivery under regional anesthesia. Additionally, data from the trauma literature have also demonstrated pulse pressure to represent an accurate surrogate of stroke volume and marker of central hypovolemia. Covertino et al. reported a direct relationship between pulse pressure and central volume reductions without any difference in mean arterial pressure. As such, pulse pressure may serve as a better maker of central hypovolemia than blood pressure alone. Therefore, pulse pressure may better predict low maternal intravascular volume and serve as a marker for post-epidural FHR changes.

Pregnancy itself is associated with alterations in blood pressure with decreased vascular tone and widening of the pulse pressure. Normal pulse pressure and variations in pregnancy are poorly described. However, in otherwise healthy non-pregnant adults, stroke volume is approximately 1.7 times the pulse pressure. Given that the stroke volume in a term pregnancy is approximated to be 100 mL/min, a normal pulse pressure in pregnancy should be approximately 60 mmHg. Therefore, a level of 45 mmHg has been proposed to define a low pulse pressure in pregnancy.

Notably, no prospective studies have evaluated a risk-factor based approach, namely the use of maternal volume status, to guide the volume of the IV fluid bolus administered prior to neuraxial anesthesia. The investigators hypothesize that in individuals with narrow pulse pressure, an increased IV fluid bolus will reduce the rate of post-epidural FHR changes. While pulse pressure variation has been best characterized as a marker of fluid responsiveness in previously healthy critically ill patients, this parameter is only readily obtained through use of an automated device (FloTrac/Vigileo system, Edwards Lifesciences, Irvine, CA) that requires an arterial line. Furthermore, pulse pressure variation has primarily been assessed in mechanically ventilated patients, which is rare in the obstetric setting. Therefore, based on the preliminary data by Miller et al., the investigators plan to use pulse pressure (and not pulse pressure variation) as a marker of intravascular volume this study with a cut point of 45 mmHg to define low pulse pressure. Given that previous studies have used IV fluid preload doses ranging from 500-1500 mL, the IV fluid dosing regimens that will be used in this study represent variations in the standard of care. A practical study design is proposed using current practice patterns for a low risk intervention in a low risk population.

Study Design:

Prospective Randomized Controlled Trial

Study Protocol:

Women meeting eligibility criteria will be recruited and randomized in a 1:1 ratio into two study groups: standard IV fluid bolus prior to epidural placement (500 mL Lactated Ringers) or "volume replacement" IV fluid bolus of 1500mL Lactated Ringers. IV fluid boluses will be infused over 30 minutes and administered within 1 hour of epidural placement. A third group will also be recruited as a control, which will include women with a pulse pressure > 45 on admission (and otherwise meet the aforementioned inclusion/exclusion criteria). The control group will receive the standard preload bolus of 500 mL prior to epidural placement.

This is a practical study using standard clinical practice methods to assess vital signs. Maternal vital signs (blood pressure, heart rate) will be collected in the left lateral recumbent position after an initial 5 minute period without activity. Automated devices will be used to assess blood pressure and pulse pressure at the following times: on admission, immediately prior to infusion of IV fluid bolus in preparation for epidural placement, immediately following IV fluid bolus infusion, at epidural test dose (T=0), every 5 minutes for 30 minutes (T=0 to T=30), and then every 10 minutes for the next 30 minutes (T=30 to T=60).

The chart will be abstracted to identify changes in the FHR and interventions. Continuous external (or internal, if placed for typical obstetric indications), fetal monitoring will be performed before and after epidural placement as is standard on our L&D unit. Treatment of hypotension with administration of vasopressors or additional IV fluid boluses along with the treatment of FHR abnormalities (maternal position changes, supplemental oxygen administration, tocolytic use, cessation of oxytocin) will be recorded. Operative delivery for non-reassuring fetal status in the 60 minutes after epidural placement will be recorded. Additionally, maternal demographic and medical/obstetric data, maternal and neonatal delivery and outcome data will be recorded.

The technique for epidural placement and dosing will be standardized as follows. Epidural dosing will consist of 5 mL of 0.125% bupivicane with 10 mcg/mL of fentanyl. This standard bolus dose will be administered and levels of sensory block and numeric patient pain scores will be recorded. If patients have not achieved a pain score of 4 or less at 15 minutes after the epidural bolus, an additional bolus will be administered to achieve appropriate pain control. The volume of additional epidural bolus will be recorded.

Two independent obstetricians blinded to the randomization group and delivery outcome will interpret the FHR tracing for one hour before and after epidural placement. The FHR tracings will be divided into 15 minute epochs and categorized using the standard ACOG categories: I, II and III. Additional information including FHR baseline, FHR variability, and the presence or absence of accelerations or decelerations will be recorded for each 15min epoch. Discrepancies between the tracing interpretations will be reviewed by a third obstetrician for development of a consensus interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy with gestational age ≥ 35 weeks
* Admission for delivery
* Age 18 or older
* Desires neuraxial analgesia in labor
* No exclusion criteria
* Maternal pulse pressure < 45 mmHg on admission (verified by repeat blood pressure)
* Category 1 FHT on admission/prior to epidural placement
* Epidural placement within 6 hours of admission to Labor and Delivery

Exclusion Criteria:

* Multiple gestation
* Intrauterine growth restriction
* Hypertensive disorders (gestational hypertension, chronic hypertension, and preeclampsia/eclampsia)
* Gestational or pregestational diabetes mellitus
* Substance abuse
* Intrauterine fetal demise
* Congenital or chromosomal fetal abnormalities
* Category II or III FHR tracing on admission to L&D (pre-epidural)
* Contraindication to neuraxial aesthesia (e.g. thrombocytopenia)
* Maternal cardiomyopathy, congenital heart disease, active pulmonary edema or any other underlying maternal cardiopulmonary condition that increases the risk of pulmonary edema
* Maternal renal insufficiency (serum creatinine > 1.0)
* Maternal hypotension (as defined in secondary outcomes below) prior to epidural placement

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin R Lappen, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Osterman MJ, Martin JA. Epidural and spinal anesthesia use during labor: 27-state reporting area, 2008. Natl Vital Stat Rep. 2011 Apr 6;59(5):1-13, 16. PMID 21553556
- [Background] Bucklin BA, Hawkins JL, Anderson JR, Ullrich FA. Obstetric anesthesia workforce survey: twenty-year update. Anesthesiology. 2005 Sep;103(3):645-53. doi: 10.1097/00000542-200509000-00030. No abstract available. PMID 16129992
- [Background] Anim-Somuah M, Smyth RM, Jones L. Epidural versus non-epidural or no analgesia in labour. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD000331. doi: 10.1002/14651858.CD000331.pub3. PMID 22161362
- [Background] Collins KM, Bevan DR, Beard RW. Fluid loading to reduce abnormalities of fetal heart rate and maternal hypotension during epidural analgesia in labour. Br Med J. 1978 Nov 25;2(6150):1460-1. doi: 10.1136/bmj.2.6150.1460. PMID 719463
- [Background] Kinsella SM, Pirlet M, Mills MS, Tuckey JP, Thomas TA. Randomized study of intravenous fluid preload before epidural analgesia during labour. Br J Anaesth. 2000 Aug;85(2):311-3. doi: 10.1093/bja/85.2.311. PMID 10992845
- [Background] Kubli M, Shennan AH, Seed PT, O'Sullivan G. A randomised controlled trial of fluid pre-loading before low dose epidural analgesia for labour. Int J Obstet Anesth. 2003 Oct;12(4):256-60. doi: 10.1016/S0959-289X(03)00071-2. PMID 15321453
- [Background] Nielsen PE, Erickson JR, Abouleish EI, Perriatt S, Sheppard C. Fetal heart rate changes after intrathecal sufentanil or epidural bupivacaine for labor analgesia: incidence and clinical significance. Anesth Analg. 1996 Oct;83(4):742-6. doi: 10.1097/00000539-199610000-00014. PMID 8831313
- [Background] Paech MJ, Godkin R, Webster S. Complications of obstetric epidural analgesia and anaesthesia: a prospective analysis of 10,995 cases. Int J Obstet Anesth. 1998 Jan;7(1):5-11. doi: 10.1016/s0959-289x(98)80021-6. PMID 15321239
- [Background] Wolfler A, Salvo I, Sortino G, Bonati F, Izzo F. Epidural analgesia with ropivacaine and sufentanil is associated with transient fetal heart rate changes. Minerva Anestesiol. 2010 May;76(5):340-5. PMID 20395896
- [Background] Hofmeyr G, Cyna A, Middleton P. Prophylactic intravenous preloading for regional analgesia in labour. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD000175. doi: 10.1002/14651858.CD000175.pub2. PMID 15494990
- [Background] Gaiser RR, McHugh M, Cheek TG, Gutsche BB. Predicting prolonged fetal heart rate deceleration following intrathecal fentanyl/bupivacaine. Int J Obstet Anesth. 2005 Jul;14(3):208-11. doi: 10.1016/j.ijoa.2004.12.010. PMID 15935647
- [Background] Nicolet J, Miller A, Kaufman I, Guertin MC, Deschamps A. Maternal factors implicated in fetal bradycardia after combined spinal epidural for labour pain. Eur J Anaesthesiol. 2008 Sep;25(9):721-5. doi: 10.1017/S0265021508004183. Epub 2008 Apr 10. PMID 18400139
- [Background] Miller NR, Cypher RL, Nielsen PE, Foglia LM. Maternal pulse pressure at admission is a risk factor for fetal heart rate changes after initial dosing of a labor epidural: a retrospective cohort study. Am J Obstet Gynecol. 2013 Oct;209(4):382.e1-8. doi: 10.1016/j.ajog.2013.05.049. Epub 2013 Jun 13. PMID 23769849
- [Background] Vricella LK, Louis JM, Mercer BM, Bolden N. Epidural-associated hypotension is more common among severely preeclamptic patients in labor. Am J Obstet Gynecol. 2012 Oct;207(4):335.e1-7. doi: 10.1016/j.ajog.2012.07.029. PMID 23021700
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Auler JO Jr, Torres ML, Cardoso MM, Tebaldi TC, Schmidt AP, Kondo MM, Zugaib M. Clinical evaluation of the flotrac/Vigileo system for continuous cardiac output monitoring in patients undergoing regional anesthesia for elective cesarean section: a pilot study. Clinics (Sao Paulo). 2010 Jun;65(8):793-8. doi: 10.1590/s1807-59322010000800009. PMID 20835557
- [Background] Convertino VA, Cooke WH, Holcomb JB. Arterial pulse pressure and its association with reduced stroke volume during progressive central hypovolemia. J Trauma. 2006 Sep;61(3):629-34. doi: 10.1097/01.ta.0000196663.34175.33. PMID 16966999
- [Background] Convertino VA, Ryan KL, Rickards CA, Salinas J, McManus JG, Cooke WH, Holcomb JB. Physiological and medical monitoring for en route care of combat casualties. J Trauma. 2008 Apr;64(4 Suppl):S342-53. doi: 10.1097/TA.0b013e31816c82f4. PMID 18385586
- [Background] Mabie WC, DiSessa TG, Crocker LG, Sibai BM, Arheart KL. A longitudinal study of cardiac output in normal human pregnancy. Am J Obstet Gynecol. 1994 Mar;170(3):849-56. doi: 10.1016/s0002-9378(94)70297-7. PMID 8141215
- [Background] Cyna AM, Andrew M, Emmett RS, Middleton P, Simmons SW. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD002251. doi: 10.1002/14651858.CD002251.pub2. PMID 17054153
- [Background] Vricella LK, Louis JM, Mercer BM, Bolden N. Impact of morbid obesity on epidural anesthesia complications in labor. Am J Obstet Gynecol. 2011 Oct;205(4):370.e1-6. doi: 10.1016/j.ajog.2011.06.085. Epub 2011 Jun 29. PMID 21864821
- [Background] ACOG Practice Bulletin No. 106: Intrapartum fetal heart rate monitoring: nomenclature, interpretation, and general management principles. Obstet Gynecol. 2009 Jul;114(1):192-202. doi: 10.1097/AOG.0b013e3181aef106. No abstract available. PMID 19546798
- [Derived] Lappen JR, Myers SA, Bolen N, Mercer BM, Chien EKS. Maternal Pulse Pressure and the Risk of Postepidural Complications: A Randomized Controlled Trial. Obstet Gynecol. 2017 Dec;130(6):1366-1376. doi: 10.1097/AOG.0000000000002326. PMID 29112650

RESULTS

PARTICIPANT FLOW:
Groups:
- Volume Replacement IV Preload: Patients in this arm will receive 1500mL of Lactated Ringer's solution
  Lactated Ringer's: IV Fluid (crystalloid) used for preload prior to epidural adminstration
Period: Overall Study
Arm/Group | Standard IV Preload | Volume Replacement IV Preload
Started | 139 | 137
Completed | 139 | 137
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard IV Preload | Volume Replacement IV Preload | Total
Number analyzed (Participants) | 139 | 137 | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 139 | 137 | 276
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (5.1) | 26.9 (5.3) | 26.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 137 | 276
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 52 | 108
  White | 65 | 62 | 127
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 20 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139 | 137 | 276

OUTCOME MEASURES:

1. Primary Outcome: Incidence of New-onset Category II or III Fetal Heart Rate Tracings
Description: Each fetal heart rate tracing was evaluated in 15 min increments from the completion of epidural placement and initial dose administration. ACOG Category I, II, and III was assigned to each 15 min increment.
Time Frame: First 60 minutes following epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | Standard IV Preload | Volume Replacement IV Preload
Number analyzed (Participants) | 139 | 137
Participants | 72 | 52

2. Secondary Outcome: New Onset Hypotension (>20% Decrease in Systolic and/or Diastolic Blood Pressure)
Time Frame: First 60 minutes following epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | Standard IV Preload | Volume Replacement IV Preload
Number analyzed (Participants) | 139 | 137
Participants | 48 | 14

3. Secondary Outcome: Interventions to Correct Maternal Hypotension or Fetal Heart Rate Abnormalities (Position Change, Supplemental Oxygen, Vasopressor Support, Emergent Operative Delivery)
Time Frame: First 60 minutes following epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | Standard IV Preload | Volume Replacement IV Preload
Number analyzed (Participants) | 139 | 137
Participants | 61 | 25

4. Secondary Outcome: Adverse Events (Pulmonary Edema)
Description: Pulmonary edema occurring after preload bolus through delivery was considered an adverse event.
Time Frame: Duration of intrapartum course
Measure: Count of Participants; unit: Participants
Arm/Group | Standard IV Preload | Volume Replacement IV Preload
Number analyzed (Participants) | 139 | 137
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard IV Preload | Volume Replacement IV Preload
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/137
Other Adverse Events (participants affected / at risk) | 0/139 | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes